CLINICAL TRIAL: NCT02835040
Title: Evaluating the Impact of a New Model of Care Designed to Improve Evidence-based Management of Community-acquired Pneumonia
Brief Title: IMPROVinG Outcomes in Community Acquired Pneumonia
Acronym: IMPROVe-GAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Health, Australia (Other Government)
Collaborators: University of Melbourne (Other); Monash University (Other); La Trobe University (Other)
Responsible Party: Principal Investigator, Melanie Lloyd, Research Coordinator, Western Health, Australia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MH 2016.014
Record Dates: First submitted 2016-05-22; First posted 2016-07-15 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Pneumonia
Keywords: Corticosteroid; Antibiotic; Early mobilization; Malnutrition
MeSH Terms: conditions — Pneumonia; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAP Service (Experimental)
  Interventions: Other: New model of service delivery
- Usual care (Active Comparator)
  Interventions: Other: Current practice

INTERVENTIONS:
Other: New model of service delivery — Introduction of a new CAP disease specific clinical team to ensure systematic implementation of standardized treatment protocols (similar to a clinical pathway) for interventions supported by Level-1 evidence.
  Arms: CAP Service
Other: Current practice — Interventions as determined by the treating General Medical team consistent with current usual practice.
  Arms: Usual care

SUMMARY:
Pneumonia is the commonest illness requiring hospitalization in Australia. Elderly patients account for most admissions and incur highest costs due to longer hospitalizations, higher readmission risks and poor functional outcomes. Previous clinical trials show a number of medical and allied health interventions can effectively shorten hospitalization or reduce readmissions, but these have been poorly and inconsistently applied in practice. This proposed research builds on previous studies by applying these interventions as a standardized combined package, evaluating their effectiveness in a "real world" Australian setting and quantifying effects on both clinical outcomes and health service costs.

DETAILED DESCRIPTION:
Each year community acquired pneumonia (CAP) causes 61,000 hospital admissions (2006-7 data) and incurs costs of more than AUD300 million in Australia. At the investigators' institution, over 1000 admissions per year have an average hospital length of stay (LOS) of 5 days and incur average clinical costs of AUD6,724 per admission (2012/13 data). Prolonged LOS not only has significant implications for organizational costs but is also strongly associated with adverse patient outcomes including loss of function due to de-conditioning and higher incidence of hospital-acquired adverse events including hospital-acquired infections, intravascular-device associated complications and antibiotic-related side effects. Reducing LOS therefore benefits both the patient and the health system. General Internal Medical (GIM) services manage the largest proportion of CAP patients at Western Health, with 47% of CAP admissions managed by GIM in 2012/13 (average age 75 with proportions with at least 1, 2 or 3 active co-morbidities 70%, 43% and 27% respectively). With population ageing, the elderly and highly multi-morbid population treated by GIM units will constitute the bulk of Australia's future health service burden for CAP.

A number of interventions for improving clinical outcomes in CAP are now supported by recently accrued level 1 evidence. Following a Cochrane review in 2011 that suggested adjunct corticosteroids accelerate time to clinical stability, a number of trials have since demonstrated favorable outcomes. Most notable are two landmark large randomized controlled trials (RCT); a study of the effect of corticosteroid on reducing treatment failure in severe CAP published in JAMA, and a study published in the Lancet in 2015 that demonstrated faster clinical recovery and shorter LOS (by 1 day) without significant adverse events.10 A subsequent meta-analysis (2000 patients from 12 RCTs) confirmed these findings and routine adjunctive corticosteroid is now widely supported though as yet not consistently deployed. Early mobilization safely and effectively reduces LOS when applied appropriately as does early switch to oral antibiotics guided by a set of well-defined basic clinical and laboratory criteria. Recently, a RCT incorporating both measures demonstrated a LOS reduction of 2 days compared to standard care. A meta-analysis of nutritional support in malnourished medical inpatients (a patient cohort that includes those admitted with CAP) showed that systematic screening for risk of malnutrition and targeted nutritional therapy intervention reduces non-elective readmission rates.

No existing study has assessed bundling all four established interventions (corticosteroid, early switch to oral antibiotics, early mobilization and systematic screening for malnutrition and targeted nutritional therapy). However, adherence to consensus guidelines for CAP is notoriously poor suggesting the major challenge will be in bridging the "evidence-practice gap" and particularly changing clinician behavior. Generalist clinicians are becoming increasingly overwhelmed by a plethora of guidelines for multiple illnesses that may co-exist in the same patient. Currently at Western Health, 43% of CAP patients receive corticosteroids, 63% physiotherapy (median time to initiation 2 days) and 65% a guideline-compliant antibiotic. No parenteral antibiotic stopping rules are in place (median 3 days). There is a current compliance rate of 72% for malnutrition risk screening in inpatients across the health service. The investigators believe therefore, that in order to address this gap between evidence and practice, an alternative service model is necessary to ensure best practice specifically for this leading contributor to health service burden.

The investigators propose evaluating a stand-alone over-arching "syndrome-based" clinical service for CAP analogous to those already applied in other areas (e.g. "stroke-services" credited with substantial improvements in outcomes from acute cerebrovascular disease). The proposed "CAP Service" would have core responsibility for ensuring comprehensive and rigorous current evidence-based best practice by application of a standardized set of management algorithms incorporating interventions supported by Level 1 evidence.

Service evaluation will take the form of a stepped wedge study design, a type of cluster RCT that is particularly well-suited to implementation and health services research. Importantly, the investigators have already successfully implemented this design in health services research at Western Health. The primary research question is to quantify the impact of a dedicated CAP Service delivering consistent and standardized evidence-based care on length of stay, costs, 30- and 90-day readmission rates and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Footscray or Sunshine Hospital meeting the standardized definition for community acquired pneumonia.

Exclusion Criteria:

* Palliated on admission.
* Enrolled in another inpatient clinical trial.

Withdrawal Criteria:

* Transferred to a non-General Medical Unit within 48-hours of admission.
* Transferred to another health service within 48-hours of admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Through study completion, an average of five days

SECONDARY OUTCOMES:
Hospital readmissions | Within 30-days and 90-days of discharge
Individual per-separation admission costing | From admission to emergency department until 90-days post-discharge
  Total cost per admission that can be directly attributed to patient inpatient stay as recorded by the Power Performance Manager software platform.
In-hospital mortality | 15 months
Proportion of patients receiving each individual evidence-based treatment recommendation | 15 months
Proportion of patients receiving all evidence-based treatment recommendations | 15-months
Incidence of hyperglycaemia in known diabetics requiring new insulin prescription | 15-months
Falls or clinical deterioration during physiotherapy | 15-months
Admission to Intensive Care Unit from medical ward during admission | 15-months
  Does not include admissions to ICU directly from the Emergency Department
Duration of mechanical ventilation and number of failed extubations | 15-months
Death within 30-days of presentation to hospital | 30-days from date of presentation to the Emergency Department
Death within 90-days of presentation to hospital | 90-days from date of presentation to the Emergency Department

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Footscray Hospital, Footscray, Victoria
  - Sunshine Hospital, St Albans, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blum CA, Nigro N, Briel M, Schuetz P, Ullmer E, Suter-Widmer I, Winzeler B, Bingisser R, Elsaesser H, Drozdov D, Arici B, Urwyler SA, Refardt J, Tarr P, Wirz S, Thomann R, Baumgartner C, Duplain H, Burki D, Zimmerli W, Rodondi N, Mueller B, Christ-Crain M. Adjunct prednisone therapy for patients with community-acquired pneumonia: a multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2015 Apr 18;385(9977):1511-8. doi: 10.1016/S0140-6736(14)62447-8. Epub 2015 Jan 19. PMID 25608756
- [Background] Mundy LM, Leet TL, Darst K, Schnitzler MA, Dunagan WC. Early mobilization of patients hospitalized with community-acquired pneumonia. Chest. 2003 Sep;124(3):883-9. doi: 10.1378/chest.124.3.883. PMID 12970012
- [Background] Carratala J, Garcia-Vidal C, Ortega L, Fernandez-Sabe N, Clemente M, Albero G, Lopez M, Castellsague X, Dorca J, Verdaguer R, Martinez-Montauti J, Manresa F, Gudiol F. Effect of a 3-step critical pathway to reduce duration of intravenous antibiotic therapy and length of stay in community-acquired pneumonia: a randomized controlled trial. Arch Intern Med. 2012 Jun 25;172(12):922-8. doi: 10.1001/archinternmed.2012.1690. PMID 22732747
- [Background] Siemieniuk RA, Meade MO, Alonso-Coello P, Briel M, Evaniew N, Prasad M, Alexander PE, Fei Y, Vandvik PO, Loeb M, Guyatt GH. Corticosteroid Therapy for Patients Hospitalized With Community-Acquired Pneumonia: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 Oct 6;163(7):519-28. doi: 10.7326/M15-0715. PMID 26258555
- [Background] Marti C, Grosgurin O, Harbarth S, Combescure C, Abbas M, Rutschmann O, Perrier A, Garin N. Adjunctive Corticotherapy for Community Acquired Pneumonia: A Systematic Review and Meta-Analysis. PLoS One. 2015 Dec 7;10(12):e0144032. doi: 10.1371/journal.pone.0144032. eCollection 2015. PMID 26641253
- [Background] Torres A, Sibila O, Ferrer M, Polverino E, Menendez R, Mensa J, Gabarrus A, Sellares J, Restrepo MI, Anzueto A, Niederman MS, Agusti C. Effect of corticosteroids on treatment failure among hospitalized patients with severe community-acquired pneumonia and high inflammatory response: a randomized clinical trial. JAMA. 2015 Feb 17;313(7):677-86. doi: 10.1001/jama.2015.88. PMID 25688779
- [Derived] Lloyd MA, Tang CY, Callander EJ, Janus ED, Karahalios A, Skinner EH, Lowe S, Karunajeewa HA. Patient-reported outcome measurement in community-acquired pneumonia: feasibility of routine application in an elderly hospitalized population. Pilot Feasibility Stud. 2019 Jul 27;5:97. doi: 10.1186/s40814-019-0481-y. eCollection 2019. PMID 31372236
- [Derived] Lloyd M, Karahalios A, Janus E, Skinner EH, Haines T, De Silva A, Lowe S, Shackell M, Ko S, Desmond L, Karunajeewa H; Improving Evidence-Based Treatment Gaps and Outcomes in Community-Acquired Pneumonia (IMPROVE-GAP) Implementation Team at Western Health. Effectiveness of a Bundled Intervention Including Adjunctive Corticosteroids on Outcomes of Hospitalized Patients With Community-Acquired Pneumonia: A Stepped-Wedge Randomized Clinical Trial. JAMA Intern Med. 2019 Aug 1;179(8):1052-1060. doi: 10.1001/jamainternmed.2019.1438. PMID 31282921
- [Derived] Skinner EH, Lloyd M, Janus E, Ong ML, Karahalios A, Haines TP, Kelly AM, Shackell M, Karunajeewa H. The IMPROVE-GAP Trial aiming to improve evidence-based management of community-acquired pneumonia: study protocol for a stepped-wedge randomised controlled trial. Trials. 2018 Feb 5;19(1):88. doi: 10.1186/s13063-017-2407-4. PMID 29402313